CLINICAL TRIAL: NCT00001860
Title: Sandostatin LAR vs. Surgery in Acromegalics With Macroadenoma
Brief Title: Sandostatin LAR Depot vs. Surgery for Treating Acromegaly
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 990162; 99-DK-0162
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2002-07

CONDITIONS: Acromegaly; Pituitary Neoplasm
Keywords: Growth Hormone; Somatostatin; Insulin-like Growth Factor-One; Acromegaly; Macroadenoma
MeSH Terms: conditions — Acromegaly; Pituitary Neoplasms

INTERVENTIONS:
Drug: Sandostatin LAR Depot versus transsphenoidal surgery

SUMMARY:
The purpose of this study is to compare the efficacy of Sandostatin LAR® (Registered Trademark) Depot to transsphenoidal surgery in previously untreated acromegalic patients with macroadenomas. The primary goal is to normalize insulin-like growth factor-1 (IGF-1) levels. Secondary goals are to compare Sandostatin LAR® (Registered Trademark) Depot treatment and transsphenoidal surgery to achieve the following goals: suppress growth hormone levels to less than or equal to 2.5 ng/mL, relieve the clinical signs and symptoms of acromegaly, reduce the size of the macroadenomas, produce few side effects, assess the prognostic value of baseline pituitary adenoma size, extension and baseline growth hormone level on post-treatment growth hormone and IGF-1 levels, and assess the resource utilization of each treatment type.

DETAILED DESCRIPTION:
The purpose of this study is to compare the efficacy of Sandostatin LAR® (Registered Trademark) Depot to transsphenoidal surgery in previously untreated acromegalic patients with macroadenomas. The primary goal is to normalize insulin-like growth factor-1 (IGF-1) levels. Secondary goals are to compare Sandostatin LAR® (Registered Trademark) Depot treatment and transsphenoidal surgery to achieve the following goals: suppress growth hormone levels to less than or equal to 2.5 ng/mL, relieve the clinical signs and symptoms of acromegaly, reduce the size of the macroadenomas, produce few side effects, assess the prognostic value of baseline pituitary adenoma size, extension and baseline growth hormone level on post-treatment growth hormone and IGF-1 levels, and assess the resource utilization of each treatment type.

ELIGIBILITY:
INCLUSION CRITERIA:

Male or female patients, 18 years of age or older.

Newly diagnosed patients with acromegaly, or previously untreated.

Presence of a pituitary tumor greater than 10 mm at greatest diameter (macroadenoma).

Lack of suppression of GH to less than 2.0 ng/mL using a regular GH RIA, or less than one ng/mL using a two-site immunoradiometric or chemiluminescent GH assay, after oral administration of 100 g of glucose.

IGF-1 levels above the upper limits of normal (adjusted for age and gender).

Demonstrated tolerance to a test dose of s.c. Sandostatin Injection.

Demonstrated responsiveness to a 100 ug s.c. Sandostatin Injection test dose, as evidenced by suppression of mean 4HR GH to less than 5 ng/mL, or to greater than 50 % of the baseline value.

Patients who are able to provide written informed consent.

EXCLUSION CRITERIA:

Patients demonstrating intolerance to a s.c. Sandostatin (octreotide acetate) test dose.

Patients who have received any prior treatment for their acromegaly, including radiotherapy, octreotide, bromocriptine, lanreotide, or prior surgery.

Female patients who are pregnant or lactating, or are of childbearing potential and not practicing a medically acceptable method of birth control.

Patients with compression of the optic chiasm significant enough to cause visual field defects on automated testing.

Patients who require surgery for relief of any neurologic signs or symptoms associated with their tumor.

Patients with symptomatic cholelithiasis.

Patients who have congestive heart failure (NYHA Class III and IV), unstable angina, sustained ventricular tachycardia, ventricular fibrillation, or a history of acute myocardial infarction within the three months preceding study entry.

Patients with liver disease such as cirrhosis, chronic active hepatitis or chronic persistent hepatitis, or persistent ALT, AST, or alkaline phosphatase 2X greater than upper limit of normal; or direct bilirubin more than 10% greater than upper limit of normal.

Patients with abnormal clinical laboratory values considered by the Investigator or the Sponsor's Medical Monitor to be clinically significant and which could affect the interpretation of the study results.

Patients who have any current or prior medical condition that may interfere with the conduct of the study or of the evaluation of its result in the opinion of the Investigator or Sponsor's Medical Monitor.

Patients who have a history of alcohol or drug abuse in the six month period prior to Visit 1.

Patients who have received any investigational drug within one month prior to Visit 1, or who plan to take an investigational drug during the study.

Patients with any mental impairment limiting their ability to comply with all study requirements.

Patients who, for any reason, will be unable to complete the entire study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5
Dates: Start 1999-08; Study Completion 2002-07

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK), Bethesda, Maryland, United States

REFERENCES:
- [Background] Barkan AL. Acromegaly. Diagnosis and therapy. Endocrinol Metab Clin North Am. 1989 Jun;18(2):277-310. PMID 2663476
- [Background] Bates AS, Van't Hoff W, Jones JM, Clayton RN. An audit of outcome of treatment in acromegaly. Q J Med. 1993 May;86(5):293-9. PMID 8327647
- [Background] Melmed S, Jackson I, Kleinberg D, Klibanski A. Current treatment guidelines for acromegaly. J Clin Endocrinol Metab. 1998 Aug;83(8):2646-52. doi: 10.1210/jcem.83.8.4995. PMID 9709926